CLINICAL TRIAL: NCT05778331
Title: The Difference Between POSEIDON Group 3 and Group 4 as Regards IVF
Acronym: POSEIDON
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MS 862/2022/2023
Record Dates: First submitted 2023-02-28; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Infertility, Female; IVF
MeSH Terms: conditions — Infertility, Female | interventions — Ovulation Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A : POSEIDON group 3: 1. Age : < 35
  2. AFC: < 5
  3. AMH : < 1.2
  4. Planning for IVF
  Interventions: Procedure: Antagonist protocol for induction of ovulation
- Group B: POSEIDON group 4: 1. Age : ≥ 35 years old
  2. AFC : < 5
  3. AMH : < 1.2
  4. Planning for IVF
  Interventions: Procedure: Antagonist protocol for induction of ovulation

INTERVENTIONS:
Procedure: Antagonist protocol for induction of ovulation — Full labs will be revised to exclude women with any chronic disease. Ultrasound to exclude any anatomical uterine problem.HSG.Women who will be categorized as Poseidon group 3 and Poseidon group 4.They will be given after that antagonist protocol with dose of HMG/FSH 300-450 I.U. per day: (Gonapure 150 I.U -follicle stimulating hormone FSH preparation of recombinant DNA technology- MinaPharm pharmaceuticals-Egypt) will be given from 2nd day of menstruation per day as starting dose then on 7th day (Cetrotide 0.25 -Cetrorelix, an anti-gonadotropin releasing hormone- MERCK SORONO-Germany) will be given daily till triggering . US will be done to evaluate follicular size from 7th day if it will be 1.8 cm or more for at least 2 follicles then (Chorimon 5000 i.u-Choriogonadotropin Alfa-IBSA-Switzerland )of total dose 10000 I.U. will be given then ovum pick up with be done after 35 h of triggering ovulation .Assessment of embryo quality

SUMMARY:
prospective observational study over POSEIDON group 3 and POSEIDON group 4 with antagonist protocol for clinical pregnancy rate outcomes

DETAILED DESCRIPTION:
Type of study: prospective observational study.

Study setting: Ain Shams University Maternity Hospital (IVF. unit) Specialized IVF centers in GIZAH

Study period: Until all needed patients have been recruited (about 6 months from start of the study).

Study population: women who attend IVF clinic who will be categorized as poor ovarian responders specifically those categorized as Poseidon group 3 and Poseidon group 4 are planning to undergo ICSI/IVF.

Sampling method: patients will be divided in 2 groups : Group A Poseidon group 3 & Group B Poseidon group 4.

Sample size: The study will be conducted on 340 patients.

Sample justification: Using PASS 15 program for sample size calculation , setting power at 80% and α-error at 0.05 , and assuming clinical pregnancy rate of 21.3% for Poseidon group 3 and 10.3% for Poseidon group 4 , sample size of 170 women per group will be needed to detect difference between groups (RK abdullah , 2020).

Ethical consideration: The study will be done after the approval of the ethical committee of the department of obstetrics and gynecology, faculty of medicine, Ain Shams University. Informed consent will be taken from all participants before recruitment in the study, and after explaining the purpose and procedures of the study. The investigator will obtain the written, signed informed consent of each subject prior to performing Specific procedures on the subject. The investigator will retain the original signed informed consent form. The study will be based on the investigator self-funding.

Study procedure:

1. Full history will be taken from targeted women (personal, previous obstetric, menstrual, surgical, previous ICSI).
2. Labs will be revised especially AMH , FSH , LH , E2 , prolactin , TSH.
3. AFC on day 2 or 3 of menses.
4. Full labs for chronic disease will be revised to exclude women with any chronic disease.
5. Ultrasound at least to exclude any anatomical uterine problem.
6. HSG .
7. Women who will be categorized as Poseidon group 3 (Group A) and Poseidon group 4 (Group B).
8. They will be given after that antagonist protocol with dose of HMG/FSH 300-450 I.U. per day: (Gonapure 150 I.U -follicle stimulating hormone FSH preparation of recombinant DNA technology- MinaPharm pharmaceuticals-Egypt) will be given from 2nd day of menstruation per day as starting dose then on 7th day (Cetrotide 0.25 -Cetrorelix, an anti-gonadotropin releasing hormone- MERCK SORONO-Germany) will be given daily till triggering . US will be done to evaluate follicular size from 7th day if it will be 1.8 cm or more for at least 2 follicles then (Chorimon 5000 i.u-Choriogonadotropin Alfa-IBSA-Switzerland )of total dose 10000 I.U. will be given then ovum pick up with be done after 35 h of triggering ovulation (B.C. Tarlatzis, 2006).
9. Assessment of embryo quality by embryologist on day 2 and day 3 to grade embryos and also checking of blastocyst formation on day 5.
10. Embryo transfer (ET) will be done when it is on day 3 or day 5 based on the number and quality of available embryos.

ELIGIBILITY:
Inclusion Criteria:

(Poseidon group 4)

1. Age : ≥ 35 years old
2. AFC : < 5
3. AMH : < 1.2
4. Planning for IVF (Poseidon group 3)

1. Age : < 35 2. AFC: < 5 3. AMH : < 1.2 4. Planning for IVF

Exclusion Criteria:

1. Chronic medical disorders such as : hypertension, diabetes, etc as it may affect embryo quality and pregnancy rate .
2. Evidence of intrauterine pathology ( polyp , fibroid , adenomyosis) as it affect implantation rate.
3. Evidence uterine congenital anomaly(septum , bicornuate ) as it affects implantation rate.
4. Evidence of hydrosalpinx as it affects implantation rate.
5. Infertility due to azoospermia (male case of infertility) as it affects the rate of fertilization.
6. Patients already on other therapies(DHEA ,steroids, etc) as it affects pregnancy rate.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: women who attend IVF clinic who will be categorized as poor ovarian responders specifically those categorized as Poseidon group 3 and Poseidon group 4 are planning to undergo ICSI/IVF.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rates. | Untill all patient has been recruited - about 6 months
  number of clinical pregnancy/ number of embryo transfer cycle for each group

SECONDARY OUTCOMES:
Implantation rate after embryo transfer | Untill all patient has been recruited - about 6 months
  number of gestational sac/ total number of transferred embryo
Number of high quality grade A embryos on day 3 and blastocyst. | Untill all patient has been recruited - about 6 months
  number of grade A embryos
Fertilization rate. | Untill all patient has been recruited - about 6 months
  number of fertilized ovum / number of retrieved oocyte

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No